CLINICAL TRIAL: NCT05018520
Title: The Safety and Effectiveness of Four Courses of R-CHOP Plus Four Courses of Rituximab Versus Six Courses of R-CHOP Plus Two Courses of Rituximab in the Treatment of Naive, Low-risk, Non-mass Diffuse Large B-cell Lymphoma: a Multi-center, Prospective, Randomized Controlled Study
Brief Title: The Safety and Effectiveness of 4R-CHOP+4R vs 6R-CHOP+2R in Newly Diagnosed Patients With DLBCL in Low Risk
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director, Hematology Department, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLK-C-2015
Record Dates: First submitted 2021-08-11; First posted 2021-08-24 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Diffuse large B cell lymphoma; Side effects; Rituximab
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4RCHOP+4R (Experimental): Four Courses of R-CHOP Plus Four Courses of Rituximab
  Interventions: Drug: Four Courses of R-CHOP Plus Four Courses of Rituximab
- 6RCHOP+2R (Experimental): Six Courses of R-CHOP Plus Two Courses of Rituximab
  Interventions: Drug: Six Courses of R-CHOP Plus Two Courses of Rituximab

INTERVENTIONS:
Drug: Six Courses of R-CHOP Plus Two Courses of Rituximab — The patients will be given RCHOP (Rituximab 375mg/m2 ivgtt, D0, Cyclophosphamide 750mg/m2, ivgtt D1, doxorubicin 50mg/m2,ivgtt D1, Vincristine 1.4mg/m2（max 2mg）, ivgtt D1 Prednisone 60mg/m2 （max 100mg）,PO,D1-D5 every 21 days for total 6 courses) followed by Rituximab (375mg/m2 d1, every 21 days for total 2 courses)
  Arms: 6RCHOP+2R
Drug: Four Courses of R-CHOP Plus Four Courses of Rituximab — The patients will be given RCHOP (Rituximab 375mg/m2 ivgtt, D0, Cyclophosphamide 750mg/m2, ivgtt D1, doxorubicin 50mg/m2,ivgtt D1, Vincristine 1.4mg/m2（max 2mg）, ivgtt D1 Prednisone 60mg/m2 （max 100mg）,PO,D1-D5 every 21 days for total 4 courses) followed by Rituximab (375mg/m2 d1, every 21 days for total 4 courses)
  Arms: 4RCHOP+4R

SUMMARY:
The Safety and Effectiveness of Four Courses of R-CHOP Plus Four Courses of Rituximab Versus Six Courses of R-CHOP Plus Two Courses of Rituximab in the Treatment of Naive, Low-risk, Non-mass Diffuse Large B-cell Lymphoma: a Multi-center, Prospective, Randomized Controlled Study

DETAILED DESCRIPTION:
Diffuse large B cell lymphoma (DLBCL) is the subtype with the highest incidence, accounting for 35.8% of B cell lymphoma. 6 to 8 cycles of R-CHOP regimen is currently the standard first-line regimen for DLBCL, however, the side effects including nausea, vomiting, neutropenia, hair loss, and heart failure can decrease the life quality and are sometimes life threatening. Recently, domestic and foreign scholars have been committed to reduce the dose of chemotherapy and improve the quality of life in low-risk patients. This study uses 4 courses of R-CHOP plus 4 courses of R (4+4 plan) versus 6 courses of R-CHOP plus 2 courses of R (6+2 plan) for the treatment of newly treated, low-risk, non-mass DLBCL patients. The promising result will create a new model for the treatment and improve the life quality of low-risk DLBCL.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed CD20 positive DLBCL based on 2016 WHO classification who achieved CR after 4 cycles of RCHOP therapy (examined by PET-CT, Deauville score 1-2)
* Treatment naïve
* IPI=0,1
* Age ≥ 14 or ≤75 years
* non-mass (The length of the lesion<7.5cm)
* ECOG=0,1
* Life expectancy>6 months
* Informed consented

Exclusion Criteria:

* Have received systemic or local treatment including chemotherapy in the past
* Have received autologous stem cell transplantation in the past
* Past medical history of other malignant tumors, except basal cell carcinoma of the skin and cervical cancer in situ
* Accompanied by uncontrolled cardiovascular and cerebrovascular diseases, coagulopathy, connective tissue diseases, severe infectious diseases and other diseases
* Primary skin, primary central nervous system lymphoma
* Left ventricular ejection fraction ≦50%
* Other concurrent and uncontrolled situation which will affect the patient's medical status based on researchers decision
* Laboratory test value during screening: (unless it is caused by lymphoma) Neutrophils <1.5*109/L Platelet<80*109/L Hemoglobin <100g/L ALT or AST is 2 times higher than the upper limit of normal, AKP and bilirubin are 1.5 times higher than the upper limit of normal E. Creatinine level is higher than 1.5 times the upper limit of normal
* Psychiatric patients or other patients who are known or suspected to be unable to fully accomplish with the research protocol
* Pregnant or lactating women
* Patients with positive HbsAg test results need to undergo HBV-DNA test and can be admitted to the group after turning negative. In addition, if the HBsAg test result is negative, but the HBcAb test is positive (regardless of the HBsAb status), HBV-DNA is also required；if the result is positive, patients also need to be treated to become negative before entering the group
* Patients living with HIV
* Patients with TP53 mutations or those who have not undergone DLBCL hot spot gene screening

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Progression of disease within 24 months | Baseline up to data cut-off (up to approximately 24 months)
  Progression of disease within 24 months was defined as the rate of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall response rate | t the end of Cycle 8 (each cycle is 21 days)
  Percentage of participants with overall response examined by PET-CT was determined on the basis of investigator assessments according to 2014 Lugano criteria
Overall survival | Baseline up to data cut-off (up to approximately 2 years)
  Overall survival was defined as the time from the date of diagnosis to the date of death from any cause. Reported is the percentage of participants with event. of disease progression or relapse, using 2014 Lugano criteria,or death from any cause, whichever occurred first.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Up to 30 days after completion of study treatment
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events
Quality of life of patients | Up to 30 days after completion of study treatment
  Quality of life of patients estimated by European organization for Research and Treatment of Cancer (EORCT) QLQ一C30 by the researchers

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No